CLINICAL TRIAL: NCT01879605
Title: Preoperative Bowel Preparation Versus no Preparation Before Spinal Surgery: a Randomised Clinical Trial
Brief Title: Study About Effect of Preoperative Bowel Preparation Versus no Bowel Preparation Before Spinal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: v57e4nbn
Record Dates: First submitted 2013-06-13; First posted 2013-06-18 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Constipation; Ileus; Surgery
Keywords: Spinal surgery; Bowel preparation; Ileus; Constipation; Well-being
MeSH Terms: conditions — Constipation; Ileus | interventions — Sorbitol; Bisacodyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Enema (Experimental): Docusate natrium and sorbitol, 240 ml enema, the evening before surgery
  Interventions: Drug: Docusate natrium and sorbitol
- Suppository (Active Comparator): Bisacodyl, suppository 10 mg, the evening before surgery.
  Interventions: Drug: Bisacodyl
- Control grup (No Intervention): No intervention

INTERVENTIONS:
Drug: Docusate natrium and sorbitol
  Other Names: Klyx
  Arms: Enema
Drug: Bisacodyl
  Other Names: Dulcolax
  Arms: Suppository

SUMMARY:
This study investigated the effect of preoperative bowel preparations for patients undergoing spinal fusion surgery.

DETAILED DESCRIPTION:
This was a randomised clinical trial with one control group and two treatment groups.

Forty-five elective spinal fusion patients were randomised into three groups who received preoperative treatment with either enema of sorbitol and docusat natrium, Bisacodyl suppository or no bowel preparation.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing spinal fusion surgery
* Age 15 years or older
* The patients had to understand oral and written Norwegian.
* Postoperative pain management via epidural catheter should have been planned.
* Exclusion Criteria:
* Constipation
* Regularly use of enema

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2007-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Defecation within 72 hours postoperatively | The study's outcome measures were recorded every evening between 17.00 and 21.00 hours

SECONDARY OUTCOMES:
Postoperative constipation | The study's outcome measures were recorded every evening between 17.00 and 21.00 hours

OTHER OUTCOMES:
The study's outcome measures were recorded every evening between 17.00 and 21.00 hours | Nausea
Pain | The study's outcome measures were recorded every evening between 17.00 and 21.00 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ida T Bjork, MNSc, PhD,, Principal Investigator — University of Oslo, Institute of Health and society
Locations (1):
- Oslo Universitetssykehus, Oslo, Oslo County, Norway